CLINICAL TRIAL: NCT04232046
Title: Efficacy of Trigger Points Massage in Severity of Chronic Tension Headache:An Unmasked, Randomized, Controlled Trial
Brief Title: Trigger Point Massage in Chronic Tension Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mazandaran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Athena Sharifi Razavi, Assistant Professor in Neurology, Mazandaran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1288
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Tension-Type Headache
Keywords: Massage; Trigger point
MeSH Terms: conditions — Tension-Type Headache | interventions — Massage

STUDY DESIGN:
Intervention Model Description: Case and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Trigger point massage
  Interventions: Other: Massage
- Control (Active Comparator): Treatment with standard drug Nortriptyline
  Interventions: Other: Massage

INTERVENTIONS:
Other: Massage — Massage the trigger points in 8 different points for 1 min in circle direction and 3 times a day.

SUMMARY:
Patients with IHS criteria of chronic tension headache , considering inclusion and exclusion criteria, enrolled to this study. They will be randomized to intervention or control group by block randomization method, then treat by standard drug( nortriptyline 10 mg daily) or trigger point massage.

They report severity, frequency, duration of headaches and number of analgesic drugs in diary during week 1 and week 4. Then data based on dairy will be analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic tension type headache according to IHS criteria
2. Finding painful trigger point in physical examination
3. no contraindication for massage
4. no prophylactic treatment
5. written inform consent

Exclusion Criteria:

1. Dementia or severe cognitive impairment
2. Under Treatment with drugs with prophylactic effect
3. History of RA or Cervicocephalic fracture or other skeletal deformity
4. Other complementary treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Headache severity change | Mean Visual Analogue Scale sore change in week 4 from the baseline
  By Visual Analogue Scale score,from 0 that indicate no pain to 10 that indicate severe pain

SECONDARY OUTCOMES:
Headache frequency change | Change in number of attacks in week 4 from the base line
  Number of attacks in week
Headache duration change | Change in Time duration in week 4 from the baseline
  Time duration ( in minutes)of attacks in week
Number of analgesic change | Change in Number of analgesic drugs used in week 4 from the baseline
  Number of analgesic drugs used during a week

IPD SHARING:
Plan to Share IPD: No